CLINICAL TRIAL: NCT02204306
Title: TSER Genotype Guided Chemotherapy in Metastatic Gastric Cancer Patients: A Phase II Study in China
Brief Title: Genotype Guided Chemotherapy in Gastric Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Yijing He, Associate Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000 Talents-CSU-GC; 1000 Plan (Other: 1000 Plan Program)
Record Dates: First submitted 2014-07-21; First posted 2014-07-30 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TSER *2/*2 *2/*3 (Other): Patients with TSER *2/*2 *2/*3 genotypes will be assigned to this group and receive standard chemotherapy contains fluorouracil. (FOLFOX 6/XELOX/SOX)
  Interventions: Genetic: TSER
- TSER*3/*3 (fluorouracil) (Other): Patients with TSER*3/*3 genotype will be randomly assigned to fluorouracil group (FOLFOX 6/XELOX/SOX) or non-fluorouracil group (DC or DO).
  Interventions: Genetic: TSER
- TSER*3/*3 (non-fluorouracil) (Other): Patients with TSER*3/*3 genotype will be randomly assigned to fluorouracil group (FOLFOX 6/XELOX/SOX) or non-fluorouracil group (DC or DO).
  Interventions: Genetic: TSER

INTERVENTIONS:
Genetic: TSER — TS gene will be genotyped for each patients prior to chemotherapy. Patients will be assigned to different arms according to specific TSER genotype.
  Other Names: TSER genotypes: *2/*2 *2/*3 *3/*3

SUMMARY:
In gastric cancer patients treated with 5-FU and cisplatin, higher tumor TS levels were associated with a less favorable response (29% vs. 68%; p=0.024). Similarly, in a study in which patients were treated with high dose 5-FU, patients with high TS expression had a response rate of only 12.5%. Conversely a response rate of 92.9% was observed in patients with low tumor TS expression. A longer but not statistically significant survival advantage was observed in patients with the TSER*2 allele compared with the TSER*3/*3 patients. Additionally, a review by Patel et al. identified approximately 20 gastric cancer studies that have found a positive association between TSER genotype and clinical response (in either direction). Therefore, the primary goal of this proposal is to prospectively genotype patients, select patients with "good risk" TSER genotypes (TSER*2*/*2 or *2/*3) and treat them with a standard 5-FU containing regimen (FOLFOX) in order to improve clinical outcomes, while randomize patients with the "poor risk" TSER genotype (*3/*3) to either the standard 5-FU containing regimen or another non-5-FU-based regimen (docetaxel/cisplatin).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed metastatic adenocarcinoma of the stomach.
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See section 9.2 for the evaluation of measurable disease.
3. No prior therapy for metastatic disease. Prior neo-adjuvant or adjuvant therapy is permitted if the disease free interval has been longer than 12 months.
4. Age between 18 and 70 years. Because no dosing or adverse event data are currently available on the use of these regimens in patients <18 years of age, children are excluded from this study.
5. Life expectancy of greater than 3 months.
6. ECOG performance status < 2 (Karnofsky >60%; see Appendix A).
7. Patients must have normal organ and marrow function as defined below:

   * Leukocytes >3,000/microliter
   * Absolute neutrophil count >1,500/microliter
   * Platelets >100,000/microliter
   * Total bilirubin < 1.5 x ULN
   * AST(SGOT)/ALT(SGPT) <2.5 x ULN if not liver metastases < 5 x ULN if known liver metastases
   * Creatinine clearance <1.5 x ULN
8. Not pregnant. Not breast feeding. If the patient or partner is of childbearing potential, the couple will use adequate birth control in accordance with local IRB policies:

   For woman of childbearing potential:

   Patient must have negative blood pregnancy test. If sexually active, woman must either be post-menopausal (over age 50 and have not had a menstrual period for one year or more, or blood FSH level in the post-menopausal range) OR agree to use appropriate contraceptive measures for the duration of the study and for 21 days after stopping study treatment. The only birth control methods for women that are acceptable for this study are: (1) surgical sterilization (previous removal of the uterus or both ovaries or a tubal ligation) OR (2) an intrauterine device (IUD), (3) double barrier methods, (4) oral contraceptives.

   For men:

   Medically acceptable contraceptives include: (1) surgical sterilization, or (2) a condom used with a spermicide. If the female partner becomes pregnant while patient is on treatment or within 21 days after stopping treatment, the study physician must be informed.
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients may not be receiving any other chemotherapy agents.
2. Patients with known active brain metastases. Patients with treated brain metastases are permitted if stable off steroids for at least 30 days. A screening head CT/MRI is not required in asymptomatic patients for this protocol.
3. History of allergic reactions to 5-FU, oxaliplatin, docetaxel, or cisplatin.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with the chemotherapies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
disease control rate | 6 and 12 weeks after the first chemotherapy
  Determine whether the disease control rate (DCR) at 6 and 12 weeks in TSER*3/*3 patients with metastatic gastric cancer will be increased by using a non fluoropyrimidine containing regimen compared to fluoropyrimidine-containing regimens.

SECONDARY OUTCOMES:
time to progression | 2 years maximum
  TTP is defined in this study as: "The length of time from the date of the start of treatment for gastric cancer until the disease starts to get worse or spread to other parts of the body."
median overall survival | 2 years maximum
  median overall survival is defined in this study as: "The length of time from the start of treatment for a disease that half of the patients in a group of patients diagnosed with the disease are still alive."

OTHER OUTCOMES:
drug toxicities | 2 years maximum
  Drug toxicities will be recorded and evaluated by NCI CTCAE v3.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Clinical Pharmacology, Changsha, Hunan, China